CLINICAL TRIAL: NCT02214277
Title: Cerebral Protection in Transcatheter Aortic Valve Replacement - The SENTINEL Study
Brief Title: Cerebral Protection in Transcatheter Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claret Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CP-10836
Record Dates: First submitted 2014-08-08; First posted 2014-08-12 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Severe Symptomatic Calcified Native Aortic Valve Stenosis
Keywords: Embolic Protection; Edwards SAPIEN THV; Edwards SAPIEN XT; TAVR; Transfemoral; Transapical; Heart Valve Diseases; Heart Diseases; TAVI; Aortic Stenosis; Aortic Valve; Transcatheter Heart Valve
MeSH Terms: conditions — Heart Valve Diseases; Heart Diseases; Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Test Arm (Experimental)
  Interventions: Device: Cerebral Protection System-The SENTINEL System with TAVR
- Control Arm (Active Comparator)
  Interventions: Device: TAVR
- Safety Arm (Other)
  Interventions: Device: Cerebral Protection System-The SENTINEL System with TAVR

INTERVENTIONS:
Device: Cerebral Protection System-The SENTINEL System with TAVR — Claret Medical Sentinel Cerebral Protection System is intended for use as an embolic protection system to contain and remove embolic material (thrombus/debris) that may enter the carotid arteries.
  Other Names: Cerebral Protection System: The SENTINEL System; TAVR Device: Edwards SAPIEN THV or Edwards SAPIEN XT
  Arms: Safety Arm; Test Arm
Device: TAVR
  Other Names: TAVR: Edwards SAPIEN THV or Edwards SAPIEN XT
  Arms: Control Arm

SUMMARY:
The Sentinel System will be a safe and effective method for capturing and removing embolic material (thrombus/debris) during transcatheter aortic valve replacement in order to reduce the ischemic burden in the cerebral anterior circulation.

DETAILED DESCRIPTION:
The Sentinel™ Cerebral Protection System is indicated for use as an embolic capture and retrieval system intended to reduce the ischemic burden in the cerebral anterior circulation while performing transcatheter aortic valve replacement.

The objective of this study is to assess the safety and efficacy of the Claret Medical Sentinel Cerebral Protection System used for embolic protection during Transcatheter Aortic Valve Replacement (TAVR) compared to TAVR standard of care (without embolic protection).

The study population is comprised of subjects with severe symptomatic calcified native aortic valve stenosis who meet the commercially approved indications for TAVR with the Edwards SAPIEN THV or SAPIEN XT and comply with the inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Approved indications for commercially available Edwards SAPIEN Transcatheter Heart Valve, model 9000TFX or SAPIEN XT, model 9300TFX meeting one of the three sub-criteria below:

   SAPIEN
   1. transfemoral delivery in subjects with severe symptomatic calcified native aortic valve stenosis without severe aortic insufficiency and with ejection fraction >20% who have been examined by a heart team including an experienced cardiac surgeon and a cardiologist and found to either be:

      1. inoperable and in whom existing co-morbidities would not preclude the expected benefit from correction of the aortic stenosis; or
      2. be operative candidates for aortic valve replacement but who have a Society of Thoracic Surgeons predicted operative risk score >8% or are judged by the heart team to be at a 15% risk of mortality for surgical aortic valve replacement.

      or
   2. transapical delivery in subjects with severe symptomatic calcified native aortic valve stenosis without severe aortic insufficiency and with ejection fraction > 20% who have been examined by a heart team including an experienced cardiac surgeon and a cardiologist and found to be operative candidates for aortic valve replacement but who have a Society of Thoracic Surgeons operative risk score 8% or are judged by the heart team to be at a 15% risk of mortality for surgical aortic valve replacement.

      SAPIEN XT (Transfemoral or Transapical only)
   3. in patients with symptomatic heart disease due to severe native calcific aortic stenosis (aortic valve area ≤ 1.0 cm2 or aortic valve area index ≤ 0.6 cm2/m2, a mean aortic valve gradient of ≥ 40 mmHg, or a peak aortic-jet velocity of ≥ 4.0 m/s), and with native anatomy appropriate for the 23, 26, or 29 mm valve system, who are judged by a heart team, including a cardiac surgeon, to be at high or greater risk for open surgical therapy (i.e., Society of Thoracic Surgeons operative risk score ≥8% or at a ≥15% risk of mortality at 30 days).
2. Compatible left common carotid artery (6.5 - 10 mm) and brachiocephalic artery (9 - 15 mm) diameters without significant stenosis (> 70%) as determined by Multi-Slice Computed Tomography (MSCT) scan or equivalent imaging modality
3. The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visit
4. The subject or the subject's legal representative has been informed of the nature of the trial, agrees to its provisions and has provided written informed consent as approved by the IRB of the respective clinical site

Exclusion Criteria:

General

1. Vasculature in the right extremity precluding 6Fr sheath radial or brachial access
2. Inadequate circulation to the right extremity as evidenced by signs of artery occlusion (modified Allen's test) or absence of radial/brachial pulse
3. Hemodialysis shunt, graft, or arterio-venous fistula involving the upper extremity vasculature
4. Evidence of an acute myocardial infarction ≤ 1 month before the intended treatment
5. Aortic valve is a congenital unicuspid or bicuspid valve; or is non-calcified
6. Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation >3+)
7. Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days of the index procedure (unless part of planned strategy for treatment of concomitant coronary artery disease)
8. Pre-existing prosthetic heart valve in any position, prosthetic ring, or severe (greater than 3+) mitral insufficiency
9. Blood dyscrasias as defined: Leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis or coagulopathy
10. Hemodynamic instability requiring inotropic support or mechanical heart assistance.
11. Need for emergency surgery for any reason
12. Hypertrophic cardiomyopathy with or without obstruction
13. Severe ventricular dysfunction with LVEF ≤20%
14. Echocardiographic evidence of intracardiac or aortic mass, thrombus, or vegetation
15. Symptomatic or asymptomatic severe occlusive carotid disease requiring concomitant CEA/stenting
16. Subject has undergone carotid stenting or carotid endarterectomy within the previous 6 weeks
17. Active peptic ulcer or upper GI bleeding within the prior 3 months
18. A known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, or clopidogrel, or sensitivity to contrast media, which cannot be adequately pre-medicated
19. Recent (within 6 months) CVA or a TIA
20. Renal insufficiency (creatinine > 3.0 mg/dL or GFR < 30) and/or renal replacement therapy at the time of screening
21. Life expectancy < 12 months due to non-cardiac co-morbid conditions
22. Subjects in whom anti-platelet and/or anticoagulant therapy is contraindicated, or who will refuse transfusion
23. Subjects who have active bacterial endocarditis or other active infections
24. Currently participating in an investigational drug or another device study
25. Subjects who have a planned treatment with any other investigational device or procedure during the study follow-up period (90 days)
26. Subject with planned concomitant surgical or transcatheter ablation for Atrial Fibrillation during the study follow-up period (90 days)
27. Any subject with a balloon valvuloplasty (BAV) within 30 days of the procedure

    Neurologic
28. Subject had active major psychiatric disease
29. Subject has severe visual, auditory, or learning impairment and who are unable to comprehend English and therefore unable to be consented for the study
30. Subjects with neurodegenerative or other progressive neurological disease or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities

    Angiographic
31. Excessive tortuosity in the right radial/brachial/subclavian artery preventing Sentinel System access and insertion
32. Subject whose brachiocephalic or left carotid artery reveals significant stenosis, calcification, ectasia, dissection, or aneurysm at the ostium or within 3 cm of the ostium

    Magnetic Resonance Imaging
33. Subject Body Mass Index (BMI) precluding imaging in scanner
34. Contraindications to MRI (subjects with any implantable temporary or permanent pacemaker or defibrillator, metal implants in field of view, metallic fragments, clips, or devices in the brain or eye before TAVR procedure)
35. Planned implantation of a pacemaker or defibrillator implantation after TAVR
36. Claustrophobia
37. Known allergy to gadolinium or contrast agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susheel Kodali, MD, Principal Investigator — Columbia University; Samir Kapadia, MD, Principal Investigator — The Cleveland Clinic
Locations (15):
- United States (14):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Houston / Memorial Hermann, Houston, Texas
  - UVA Advanced Cardiac Valve Center, Charlottesville, Virginia
  - UW Medical Center, Seattle, Washington
- Herzzentrum Leipzig - Universitatsklinik, Leipzig, Germany

REFERENCES:
- [Result] Kapadia SR, Kodali S, Makkar R, Mehran R, Lazar RM, Zivadinov R, Dwyer MG, Jilaihawi H, Virmani R, Anwaruddin S, Thourani VH, Nazif T, Mangner N, Woitek F, Krishnaswamy A, Mick S, Chakravarty T, Nakamura M, McCabe JM, Satler L, Zajarias A, Szeto WY, Svensson L, Alu MC, White RM, Kraemer C, Parhizgar A, Leon MB, Linke A; SENTINEL Trial Investigators. Protection Against Cerebral Embolism During Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2017 Jan 31;69(4):367-377. doi: 10.1016/j.jacc.2016.10.023. Epub 2016 Nov 1. PMID 27815101
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/27815101

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety Arm: Safety Arm patients received TAVR and the Sentinel System. Patients enrolled in this arm of the study received safety follow-up at discharge, at 30 days and 90 days post-procedure; and neurological evaluation at baseline, discharge, 30 days and 90 days (only in the case of a stroke ≤ 30 days) post procedure. Safety Arm patients did not receive MRI.
  The Safety Arm was combined with the Test Arm for analysis of safety endpoints.
- Test Arm: Test Arm patients received TAVR and the Sentinel System. Patients enrolled in this arm of the study underwent safety follow-up at discharge, at 30 and at 90 days post-procedure; MRI assessment for efficacy at baseline, 2-7 days and 30 days post-procedure; neurological evaluation at baseline, discharge, 30 days and 90 days (only in the case of a stroke ≤ 30 days) post procedure; neurocognitive evaluation at baseline, 2-7 days (optional), 30 days and 90 days post-procedure; Quality of Life assessment at baseline, 30 days and 90 days; and histopathological evaluation of debris captured in the Sentinel device filters.
  The Test Arm was compared to the Control Arm for analysis of MRI related endpoints, and was combined with the Safety Arm for analysis of safety endpoints.
- Control Arm: Control Arm patients received TAVR only. Patients enrolled in this arm of the study underwent safety follow-up at discharge, at 30 and at 90 days post-procedure; MRI assessment for efficacy at baseline, 2-7 days and 30 days post-procedure; neurological evaluation at baseline, discharge, 30 days and 90 days (only in the case of a stroke ≤ 30 days) post procedure; neurocognitive evaluation at baseline, 2-7 days (optional), 30 days and 90 days post-procedure; and Quality of Life assessment at baseline, 30 days and 90 days.
  The Control Arm was compared to the Test arm for MRI related endpoints.
Period: Overall Study
Arm/Group | Safety Arm | Test Arm | Control Arm
Started | 123 | 121 | 119
Completed | 104 | 96 | 85
Not Completed | 19 | 25 | 34

BASELINE CHARACTERISTICS:
Groups:
- Safety Arm: Safety Arm patients received TAVR and the Sentinel System. Patients enrolled in this arm of the study received safety follow-up at discharge, at 30 days and 90 days post-procedure; and neurological evaluation at baseline, discharge, 30 days and 90 days (only in the case of a stroke ≤ 30 days) post procedure.
- Test Arm: Test Arm patients received TAVR and the Sentinel System. Patients enrolled in this arm of the study underwent safety follow-up at discharge, at 30 and at 90 days post-procedure; MRI assessment for efficacy at baseline, 2-7 days and 30 days post-procedure; neurological evaluation at baseline, discharge, 30 days and 90 days (only in the case of a stroke ≤ 30 days) post procedure; neurocognitive evaluation at baseline, 2-7 days (optional), 30 days and 90 days post-procedure; Quality of Life assessment at baseline, 30 days and 90 days; and histopathological evaluation of debris captured in the Sentinel device filters.
- Control Arm: Control Arm patients received TAVR only. Patients enrolled in this arm of the study underwent safety follow-up at discharge, at 30 and at 90 days post-procedure; MRI assessment for efficacy at baseline, 2-7 days and 30 days post-procedure; neurological evaluation at baseline, discharge, 30 days and 90 days (only in the case of a stroke ≤ 30 days) post procedure; neurocognitive evaluation at baseline, 2-7 days (optional), 30 days and 90 days post-procedure; and Quality of Life assessment at baseline, 30 days and 90 days.
- Total: Total of all reporting groups
Arm/Group | Safety Arm | Test Arm | Control Arm | Total
Number analyzed (Participants) | 123 | 121 | 119 | 363
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.5 (8.98) | 82.0 (7.95) | 83.4 (7.90) | 82.3 (8.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 63 | 58 | 189
  Male | 55 | 58 | 61 | 174
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 1 | 4
  Not Hispanic or Latino | 123 | 118 | 118 | 359
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 1 | 1 | 10
  White | 109 | 115 | 115 | 339
  More than one race | 1 | 2 | 2 | 5
  Unknown or Not Reported | 3 | 2 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 98 | 95 | 96 | 289
  Germany | 25 | 26 | 23 | 74
STS PROM Score [Mean (Standard Deviation); unit: units on a scale] — The Society of Thoracic Surgeons' (STS) predicted risk of mortality (PROM) score is used to predict the risk of operative mortality and morbidity of surgery. It is based on patient demographic and clinical variables, and scores are divided into four categories: low risk (<4%),intermediate risk (>=4% to <8%), high risk (>=8% to <12%) ,very high risk (>=12%).
  units on a scale | 6.2 (3.17) | 6.4 (3.28) | 7.5 (4.66) | 6.7 (3.79)
History of Atrial Fibrillation [Count of Participants; unit: Participants] | 37 | 42 | 36 | 115

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Median Total New Lesion Volume in Protected Territories Between Test and Control Arms as Assessed by DW-MRI at Day 2-7 Post-procedure.
Description: Total new lesion volume is defined as the sum of all diffusion-positive new cerebral lesions in post-TAVR DW-MRI relative to the pre-TAVR DW-MRI scans. Protected territories are defined as brain territories uniquely perfused by the vessels protected by the Sentinel System, namely the left and right carotid arteries, and the right vertebral artery.
Time Frame: Day 2-7 Post-Procedure
Population: ITT with Imputation. Test Arm compared to the Control Arm.
Measure: Median (Inter-Quartile Range); unit: mm3
Groups:
- Test Arm: Test Arm patients received TAVR and the Sentinel System. Patients enrolled in this arm of the study underwent safety followup at discharge, at 30 and at 90 days postprocedure; MRI assessment for efficacy at baseline, 2-7 days and 30 days postprocedure; neurological evaluation at baseline, discharge, 30 days and 90 days (only in the case of a stroke ≤ 30 days) post procedure; neurocognitive evaluation at baseline, 2-7 days (optional), 30 days and 90 days postprocedure; Quality of Life assessment at baseline, 30 days and 90 days; and histopathological evaluation of debris captured in the Sentinel device filters.
Arm/Group | Test Arm | Control Arm
Number analyzed (Participants) | 121 | 119
mm3 | 109.1 [36.9 to 379.7] | 174 [39.6 to 469.3]

2. Primary Outcome: Patients With Major Adverse Cardiac and Cerebrovascular Events (MACCE) at 30 Days
Description: Primary Safety Endpoint: MACCE (all death, all stroke, and acute kidney injury class 3 within 72 hours or discharge, whatever occurs first) at 30 days compared to a historical performance goal of 18.3%.
Time Frame: 30 Days Post-Procedure
Population: Safety Arm and Test Arm. ITT with imputation.
Measure: Count of Participants; unit: Participants
Groups:
- Safety Cohort: The Safety Cohort is the combination of the Safety and Test Arms.
Arm/Group | Safety Cohort
Number analyzed (Participants) | 244
Participants | 18

3. Secondary Outcome: Captured Debris Histopathology (Observational)
Time Frame: Post-procedure
Population: Only Test Arm patients had debris samples collected. Only samples with evaluable filters were used in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Arm
Number analyzed (Participants) | 105
Participants
  Debris present | 104
  No debris present | 1

ADVERSE EVENTS:
Time Frame: 0-30 days
Groups:
- Safety Cohort (Test + Safety Arms): The Safety Cohort is the combination of the Safety and Test Arms. Patients enrolled in these arms of the study underwent safety follow-up at discharge, at 30 and at 90 days post-procedure.
- Control Arm: Control Arm patients received TAVR only. Patients enrolled in this arm of the study underwent safety follow-up at discharge, at 30 and at 90 days post-procedure.
Arm/Group | Safety Cohort (Test + Safety Arms) | Control Arm
All-Cause Mortality (participants affected / at risk) | 11/244 | 4/119
Serious Adverse Events (participants affected / at risk) | 17/244 | 11/119
Other Adverse Events (participants affected / at risk) | 158/244 | 79/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Cohort (Test + Safety Arms) (N=244) | Control Arm (N=119)
Death (Cardiac disorders) | 3 (3) | 2 (2)
Stroke (Nervous system disorders) | 13 (13) | 10 (10)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Cohort (Test + Safety Arms) (N=244) | Control Arm (N=119)
Abnormal Lab Value (General disorders) | 15 (18) | 8 (9)
Access Site Hematoma (Injury, poisoning and procedural complications) | 13 (13) | 6 (6) — All vascular access sites , including Sentinel (radial, brachial) and TAVR access
Anemia (Blood and lymphatic system disorders) | 23 (24) | 11 (11)
Arrhythmia (Cardiac disorders) | 13 (14) | 10 (10)
Cardiac Arrest (Cardiac disorders) | 4 (4) | 6 (6)
Bleed, Operative or Post-Operative (General disorders) | 12 (13) | 6 (6)
Conduction System Injury (Cardiac disorders) | 42 (47) | 30 (36)
Fever (General disorders) | 15 (15) | 3 (3)
Hypertension (General disorders) | 11 (11) | 9 (9)
Neurological Event, Imaging Only (Nervous system disorders) | 30 (31) | 23 (24)
Other (General disorders) | 53 (74) | 30 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No